CLINICAL TRIAL: NCT06044896
Title: Physiological Effects of Lateral Body Positioning on Regional Ventilation and Ultrasound Diaphragmatic Mobility in Healthy Subjects: an Experimental Study
Brief Title: Physiology of Body Lateralization on Regional Lung Ventilation Study
Acronym: LATLUNGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other); Coordination for the Improvement of Higher Education Personnel (Other); Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Shirley Lima Campos, Principal Researcher, University of Pernambuco
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: UFPE 5.980.254
Record Dates: First submitted 2023-08-30; First posted 2023-09-21 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Healthy Individuals
Keywords: Healthy Volunteers; Patient Positioning; Pulmonary Ventilation
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine Positioning (Experimental): The participant will be in the supine position.
  Interventions: Procedure: Supine Positioning
- Body Lateral Positioning (Experimental): The participant will be in the body lateral position at 30 degrees.
  Interventions: Procedure: Body Lateral Positioning

INTERVENTIONS:
Procedure: Supine Positioning — The participant will be guided to the Multicare bed and will be positioned supine with the headboard not tilted. At this point, the participant will already have the EIT electrode belt and head, trunk and lower limb cushions around it, providing stability. After the participant has been correctly positioned, ventilatory monitoring will begin using the EIT. The environment must be fully controlled, that is, with adequate lighting, all collection members in silence, as well as the devices in the place, air-conditioned environment, without exposing the participant to heat or cold. Before starting the collection, the volunteer will be asked to try not to sleep or talk, making it clear that any discomfort can be reported at any time. To keep the volunteer awake, visual and sound stimuli can be performed. Furthermore, if you cough or sigh, the collection will restart. The intervention will last 5 minutes and will be repeated twice, with intervals between body lateralization.
  Other Names: Supine Position; Supine
  Arms: Supine Positioning
Procedure: Body Lateral Positioning — The participant will start from the bench press to the 30-degree lateral position. The cushions placed at the beginning of the collection will provide stability so that the inclination does not compromise the correct positioning of the participant, preventing them from sliding on the bed. Furthermore, it is also a safety measure for the participant. The environment will be controlled throughout the intervention and visual and sound effects will also be performed in lateral positioning. The volunteer will remain in this position for five minutes and shortly after will be placed in the supine position again. To start the protocol for the second and final time, the participant will have a washout time of thirty minutes.
  Other Names: Automatic patient positioning; Continuous lateral rotation therapy; Lateral rotation therapy; Continuous rotational therapy; Kinetic bed therapy; Lateral change Positioning; Automated lateral rotation; Rotating bed; Automatic lateral therapy
  Arms: Body Lateral Positioning

SUMMARY:
The goal of this experimental study, with crossover design, is to analyze the effects of body lateralization applied at 30 degrees compared to the supine position on the distribution of ventilation and regional lung aeration in healthy individuals.

The main study questions to be answered are:

* Question 1: What are the immediate effects of 30 degree body lateralization on the distribution of regional ventilation and lung aeration in healthy individuals?
* Question 2: What is the effect of body lateralization on diaphragmatic mobility in the dependent or non-dependent hemithorax?

Participants will be submitted to changes in positioning in bed, considering a randomized sequence of interventions, between supine position and body lateralization at 30 degrees, using the Multicare bed (Linet, Czech Republic). The interventions were repeated twice each with a 30-minute washout in each sequence.

Participants will perform assessment of lung function and respiratory muscle strength with the instruments:

* Manovacuometry
* Spirometry
* Ventilometry
* Respiratory Diagnostic Assistant

The supine and body lateralization positions will be compared, with the primary outcomes being lung aeration and ventilation distribution assessed using Electrical Impedance Tomography. The secondary outcome will be diaphragmatic mobility measured through lung ultrasound.

Groups:

* Supine position
* Body lateralization

Effects

* Lung aeration
* Distribution of ventilation
* Diaphragmatic mobility

DETAILED DESCRIPTION:
Body positioning is a therapy used in the hospital environment to improve oxygenation. Recent studies recommend lateralization therapy to improve lung function locally by positioning the chest region of interest upwards. However, there are still gaps in the description of the effects of body lateralization on lung aeration and ventilation between non-dependent and gravity-dependent regions and on diaphragmatic mobility.

The objective of this study is to analyze the acute effects of lateralization on the aeration and distribution of lung ventilation, in comparison with the supine position, in healthy subjects. In addition, the effect of body positioning on diaphragm kinetics was evaluated.

This is a crossover study, which will be carried out at the Hospital das Clínicas of the Federal University of Pernambuco (HC-UFPE). The sample will consist of 30 healthy volunteers, aged between 18 and 59 years, of both sexes.

The change of body position will be performed using the Multicare bed (Linet, Praga,Czech Republic).

Lung ventilation and aeration will be evaluated with an Enlight 1800 electrical impedance tomography (EIT) (Timpel Medical, São Paulo, Brazil). The EIT images will be segmented into four regions of interest (ROIs: anterior right, anterior left, posterior right and posterior left. Diaphragm mobility will be quantified by diaphragmatic ultrasound in the supine and lateral positions.

The study was approved by the Research Ethics Committee of the Hospital das Clínicas of the Federal University of Pernambuco (EBSERH), in accordance with the norms of the National Health Council (Resolution 466/12) for research in human beings (opinion number 5,980.254).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Volunteers aged between 18 and 59 years old (youth/adults)
* Volunteers of both sexes

Exclusion Criteria:

* Individuals with contraindications for the use of manovacuometry, spirometry, ventilometry will be excluded
* Volunteers who did not tolerate the positioning or interventions
* Individuals with Grade III obesity (BMI > 40)
* Participants with below-normal prediction values for manovacuometry and spirometry according to predefined formulas for men and women
* History of flu syndrome in the last seven days.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Change in end-expiratory lung impedance (Delta EELZ) | Not later than 12 months after primary completion date
  Lung aeration will be assessed using Electrical Impedance Tomography (EIT). Regional EELZ will be calculated and analyzed concerning intervention times.
  The change in aeration distribution or change in end-expiratory lung impedance (Delta EELZ) will be determined by comparing pre- and post-intervention EELZ for lung quadrants and dependent/non-dependent regions in each intervention.
  End-expiratory lung impedance (EELZ) represents the sum of the end-expiratory impedance values of the pixels in a given region of interest. Regions of interest include: right anterior, left anterior, right posterior and left posterior, and functionally, dependent or non-dependent lung.
  Continuous EIT monitoring will occur, and outcomes will be assessed before and after each intervention, each lasting five minutes.
  Data are given in:
  * arbitrary units (a.u.)
  * mililiters
  * percentages
Change in distribution of lung ventilation (Delta Z) | Not later than 12 months after primary completion date
  The distribution of lung ventilation will also be assessed using electrical impedance tomography.
  The impedance variation (Delta Z) represents the sum of the impedance values of the pixels in a given region of interest. Regions of interest include: right anterior, left anterior, right posterior and left posterior, and functionally, dependent or non-dependent lung.
  The change in distribution of lung ventilation will be obtained by the difference between the Delta Z before and after each intervention, comparing the measurements of the lung quadrants and in the dependent and non-dependent lung regions for each intervention.
  Continuous EIT monitoring will occur, and outcomes will be assessed before and after each intervention, each lasting five minutes.
  Data are given in:
  * arbitrary units (a.u.)
  * mililiters
  * percentages

SECONDARY OUTCOMES:
Difference in diaphragmatic mobility measured by ultrasound between the supine and body lateralization positions. | Not later than 12 months after primary completion date
  Diaphragmatic mobility will be evaluated in the supine position and in the body lateralization position during the intervention using ultrasound, according to protocol from TESTA, A. et al 2011.
  Measurements will be carried out with the patient breathing spontaneously in supine and body lateralization position at 30º.
  Data are given in:
  • Millimeters.

OTHER OUTCOMES:
Respiratory pattern variables | Not later than 12 months after primary completion date
  Respiratory pattern variables will be measured by the Respiratory Diagnostic Assistant.
  The algorithm of the "Respiratory Diagnostic Assistant" device relates the variables respiratory rate, tidal volume, minute volume, inspiratory flow, expiratory flow, relationship between inspiratory and expiratory times.
  Data are given in:
  * Respiratory rate in incursion per minute
  * Tidal volume (measured in liters)
  * Minute volume (measured in liters);
  * Inspiratory flow (measured in liters);
  * Expiratory flow (measured in liters);
  * Ti/Ttotal, (measured in seconds)
  * I:E, relationship between inspiratory and expiratory times
  * Volume vs time;
  * Flow vs time.
Frequency of normal and altered breathing patterns | Not later than 12 months after primary completion date
  The frequency of normal and altered breathing patterns will be measured by the Respiratory Diagnostic Assistant.
  The "Respiratory Diagnosis Assistant" algorithm provides the classification of the diagnosis of breathing patterns as normal or altered, considering the input variables of flow, volume and time.
  * The normal breathing pattern described in the frequency of cases is when there is no change assessed by the algorithm.
  * The altered breathing pattern described in the frequency of cases are changes in the breathing pattern variables captured by the device's flow sensor during breathing at rest.
  Data are given in:
  • Absolut and relative frequencies
Lung function measured by Spirometry | Not later than 12 months after primary completion date
  Lung function tests are performed by the callibrated spirometer following American Thoracic Society guidelines (2019).
  The analysis variables will be:
  * Forced vital capacity (FVC) - given in liters and percentage of predicted value
  * Forced expiratory volume in 1 second - (FEV1) - given in liters and percentage of predicted value
  * Relationship between FVC/FEV1 - given in measured value and percentage of predicted value
  Furthermore, it allows you to draw up a functional diagnosis:
  * Normal
  * Obstructive ventilatory disorder (mild, moderate or severe)
  * Restrictive ventilatory disorder (mild, moderate or severe)
  * Mixed ventilatory disorder (with detection of obstructive and restrictive abnormality) Data are given in: Percentages
Lung volumes at rest breathing | Not later than 12 months after primary completion date
  Lung volumes at rest breathing will be measured by calibrated ventilometer (Ferraris Mark 8 Wright Respirometer®,. United Kingdom).
  Tidal volume (Vt) will be obtained by the ratio between minute volume (MV) and the respiratory rate (RR) observed during one minute of breathing at rest (Vt = MV/RR)
  Data are given in:
  * Minute volume (MV) measured in liters per minute;
  * Tidal volume (TV), measured in liters.
Lung capacities | Not later than 12 months after primary completion date
  Lung capacities will be measured by calibrated ventilometer (Ferraris Mark 8 Wright Respirometer®,. United Kingdom).
  Inspiratory capacity (IC) - It's the maximum volume voluntarily inspired from the end of a spontaneous expiration (from the resting expiratory level).
  Slow vital capacity (SVC) - measurement taken slowly, starting from a position of full inspiration for complete exhalation.
  Data are given in:
  * Inspiratory capacity - measured in liters
  * Slow vital capacity - measured in liters
Maximum inspiratory pressure (MIP) | Not later than 12 months after primary completion date
  Measurement of the maximum static inspiratory pressure that a subject can generate at the mouth measuring inspiratory muscle strength measured by digital manometer (MVD300u, Homed, Brazil)
  * Maximum inspiratory pressure (measured in cmH2O)
  * Maximum predicted inspiratory pressure (predicted %) - MIP predicted =63,27-0,55 (age)+17,96 (sex)+0,58 (weight )
  Data are given in:
  * CmH2O
  * percentage of predicted value
Maximum expiratory pressure (MEP) | Not later than 12 months after primary completion date
  Measurement of the maximum static expiratory pressure that a subject can generate at the mouth measuring expiratory muscle strength measured by digital manometer (MVD300u, Homed, Brazil)
  * Maximum expiratory pressure (cmH2O)
  * Maximum predicted expiratory pressure (predicted %)
  MEP =-61,41+2,29 (age)-0,03 age2)+33,72 (sex)+1,40 (waist)
  Data are given in:
  * CmH2O
  * percentage of predicted value

CONTACTS AND LOCATIONS:
Overall Officials: Layane Santana, Study Director — University of Pernambuco; Shirley Campos, Principal Investigator — University of Pernambuco
Locations (2):
- Brazil (2):
  - Shirley Campos, Recife, Pernambuco
  - Hospital das Clínicas da UFPE, Recife

IPD SHARING:
Plan to Share IPD: Yes
Participant characteristics Medical history Clinical measurements Functional results Images (USG) Adverse events
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Through study completion, an average of 1 year.
Access Criteria: Individual participant data (IPD) access will be granted by the PI after request review for approval via email. It will be shared with researchers and general public of interest on the subject for descriptive analyses related to our sample. A committee of researchers will be in charge of discussing the request before approving the access.

REFERENCES:
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Testa A, Soldati G, Giannuzzi R, Berardi S, Portale G, Gentiloni Silveri N. Ultrasound M-mode assessment of diaphragmatic kinetics by anterior transverse scanning in healthy subjects. Ultrasound Med Biol. 2011 Jan;37(1):44-52. doi: 10.1016/j.ultrasmedbio.2010.10.004. PMID 21144957
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Derived] Costa LSP, Reinaux CMA, Junior EFFS, Leite WS, Brandao DC, de Andrade AD, Roldan R, Morais CCA, Campos SL. Physiology of body lateralization on regional lung ventilation and lung volumes in healthy subjects: Within-subjects design. PLoS One. 2025 Oct 30;20(10):e0335622. doi: 10.1371/journal.pone.0335622. eCollection 2025. PMID 41166369